CLINICAL TRIAL: NCT00301145
Title: Treatment of Nicotine Dependence in a Health Care Setting
Brief Title: Varenicline Tartrate With Telephone-Based Counseling and/or Internet-Based Counseling in Helping Adults Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SRI International (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000455745; SRI-751
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Varenicline; Counseling

INTERVENTIONS:
Behavioral: smoking cessation intervention
Drug: varenicline
Other: counseling intervention
Other: internet-based intervention

SUMMARY:
RATIONALE: Varenicline tartrate may help people quit smoking by decreasing the symptoms of nicotine withdrawal. It is not yet known whether varenicline tartrate is more effective in helping people stop smoking when given together with a telephone-based counseling program, and Internet-based counseling program, or both programs.

PURPOSE: This randomized clinical trial is studying how well giving varenicline tartrate together with a telephone-based counseling program and/or an Internet-based counseling program works in helping adults stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of varenicline with telephone counseling vs Internet-based counseling vs telephone counseling and Internet-based smoking cessation interventions in adult smokers.
* Determine individual or group differences in patients undergoing these interventions.
* Determine heterogeneity in responsiveness in regard to the Classification and Regression Tree Analysis in patients undergoing these interventions.
* Determine the effectiveness of these interventions in regard to recruitment, implementation, barriers to treatment, exposure to intervention, satisfaction with treatment, treatment contamination, and program maintenance.
* Determine the cost-effectiveness of these interventions.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 3 intervention arms.

* Arm I: Patients undergo a proactive telephone-based (PTB) smoking cessation program.
* Arm II: Patients undergo a web-based (WB) smoking cessation program.
* Arm III: Patients undergo an integrated PTB/WB smoking cessation program. Beginning 1 week before the target quit date, all patients receive oral varenicline once daily for 3 days and then twice daily for up to 12 weeks. They also receive a mailed packet containing a welcome letter, description of the intervention services offered, a privacy notice, a Free & Clear Quit Kit (comprehensive education/self-help materials including health smoking substitutions), a phone call to orient the patient to the intervention to which they are randomized, and access to a toll-free support line. All patients undergo a pre-treatment assessment (pre-quit) and 3 post-quit assessments at 21 days, 12 weeks, and 6 months after their original scheduled quit date to determine medication adherence, treatment utilization, point-prevalent smoking outcomes, and continuous nonsmoking.

PROJECTED ACCRUAL: A total of 1,200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Smokes 10 or more cigarettes/day over the past year AND ≥ 5 cigarettes/day within the past week
* Planning to stop smoking in 4-6 weeks
* Member of Group Health Cooperative (GHC) and planning to stay enrolled for the next 6 months
* Eligible for the Free & Clear program
* Enrolled in the COMPASS study using bupropion hydrochloride medication
* No prior participation in GHC's Free & Clear smoking cessation program within the past 6 months

PATIENT CHARACTERISTICS:

* In good general health
* Sufficient verbal and written English
* Dependable access to a telephone and the Internet
* Not currently drinking ≥ 14 alcoholic drinks per week and/or binge drinking ≥ 2 times in the past month
* Not pregnant or nursing
* No plan to become pregnant
* No severe chronic heart disease (e.g, myocardial infarction within the past 3 months)
* No severe chronic obstructive pulmonary disease that ever required hospitalization or oxygen treatment
* No diagnosis of or treatment for a psychotic disorder (e.g., schizophrenia, bipolar disorder, or mania)
* Not having certain kidney problems

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent use of medications contraindicated with bupropion hydrochloride or known to lower seizure threshold (e.g., antidepressant, antipsychotic, monamine oxidase inhibitor, or protease inhibitor)
* No concurrent use of recreational or street drugs
* No concurrent use of bupropion hydrochloride or nicotine replacement therapy
* No concurrent cimetidine, metformin, phenformin, pindolol, procainamide
* Not on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E. Swan, PhD, Study Chair — SRI International
Locations (3):
- United States (3):
  - SRI International, Menlo Park, California
  - Center for Health Studies, Seattle, Washington
  - Free & Clear, Incorporated, Seattle, Washington

REFERENCES:
- [Result] Nishita DM, Jack LM, McElroy M, McClure JB, Richards J, Swan GE, Bergen AW. Clinical trial participant characteristics and saliva and DNA metrics. BMC Med Res Methodol. 2009 Oct 29;9:71. doi: 10.1186/1471-2288-9-71. PMID 19874586
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Swan GE, Javitz HS, Jack LM, Wessel J, Michel M, Hinds DA, Stokowksi RP, McClure JB, Catz SL, Richards J, Zbikowski SM, Deprey M, McAfee T, Conti DV, Bergen AW. Varenicline for smoking cessation: nausea severity and variation in nicotinic receptor genes. Pharmacogenomics J. 2012 Aug;12(4):349-58. doi: 10.1038/tpj.2011.19. Epub 2011 May 24. PMID 21606948
- [Derived] Catz SL, Jack LM, McClure JB, Javitz HS, Deprey M, Zbikowski SM, McAfee T, Richards J, Swan GE. Adherence to varenicline in the COMPASS smoking cessation intervention trial. Nicotine Tob Res. 2011 May;13(5):361-8. doi: 10.1093/ntr/ntr003. Epub 2011 Feb 24. PMID 21350041
- [Derived] Zbikowski SM, Jack LM, McClure JB, Deprey M, Javitz HS, McAfee TA, Catz SL, Richards J, Bush T, Swan GE. Utilization of services in a randomized trial testing phone- and web-based interventions for smoking cessation. Nicotine Tob Res. 2011 May;13(5):319-27. doi: 10.1093/ntr/ntq257. Epub 2011 Jan 31. PMID 21330267
- [Derived] McClure JB, Swan GE, Catz SL, Jack L, Javitz H, McAfee T, Deprey M, Richards J, Zbikowski SM. Smoking outcome by psychiatric history after behavioral and varenicline treatment. J Subst Abuse Treat. 2010 Jun;38(4):394-402. doi: 10.1016/j.jsat.2010.03.007. Epub 2010 Apr 2. PMID 20363092
- [Derived] McClure JB, Swan GE, Jack L, Catz SL, Zbikowski SM, McAfee TA, Deprey M, Richards J, Javitz H. Mood, side-effects and smoking outcomes among persons with and without probable lifetime depression taking varenicline. J Gen Intern Med. 2009 May;24(5):563-9. doi: 10.1007/s11606-009-0926-8. Epub 2009 Feb 24. PMID 19238488
- [Derived] Halperin AC, McAfee TA, Jack LM, Catz SL, McClure JB, Deprey TM, Richards J, Zbikowski SM, Swan GE. Impact of symptoms experienced by varenicline users on tobacco treatment in a real world setting. J Subst Abuse Treat. 2009 Jun;36(4):428-34. doi: 10.1016/j.jsat.2008.09.001. Epub 2008 Nov 11. PMID 19004600